CLINICAL TRIAL: NCT04830111
Title: The Effect of Heart Rate Variability Biofeedback Training on the Physical and Mental Health of Intrapartum Women
Brief Title: The Effect of Heart Rate Variability Biofeedback Training on Health of Intrapartum Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taipei University of Nursing and Health Sciences (Other)
Responsible Party: Principal Investigator, Wan-Lin Pan, assistant professor, National Taipei University of Nursing and Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 109-E-11
Record Dates: First submitted 2021-03-16; First posted 2021-04-02 (Actual); Last update posted 2024-01-26 (Actual); Status verified 2024-01

CONDITIONS: Mental Stress
MeSH Terms: conditions — Stress, Psychological

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- heart rate variability biofeedback training group (Experimental): The goal of heart rate variability biofeedback is to increase heart rate variability through paced breathing exercises, which have shown to be effective in reducing stress and anxiety in general adult populations.
  Interventions: Device: heart rate variability biofeedback Application (Eureka iDestressor)
- Care as usual (No Intervention): In this condition, all of this group take care by hospital routine and the questionnaires were completed over a period with similar intervals.

INTERVENTIONS:
Device: heart rate variability biofeedback Application (Eureka iDestressor) — heart rate variability biofeedback protocol duration time is 10 min twice/day for 5days
  Arms: heart rate variability biofeedback training group

SUMMARY:
In this study, the investigators examined the efficacy of heart rate variability biofeedback on physical and mental health problems in childbirth women.

DETAILED DESCRIPTION:
In this study, the investigators examined the efficacy of heart rate variability biofeedback on physical and mental health problems in childbirth women. The following validated self-report measures were administered before and at five days after the intervention, Perceived stress scale-10, Beck Anxiety Inventory, and Edinburgh Postnatal Depression Scale.

ELIGIBILITY:
Inclusion Criteria:

* woman
* aged 20 years or more
* able to understand and write Chinese
* singleton birth
* having a full-term and healthy newborn

Exclusion Criteria:

* suicidal ideations
* psychosis
* medical or obstetric complications

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 82 (Actual)
Dates: Start 2020-08-12 (Actual); Primary Completion 2022-03-02 (Actual); Study Completion 2022-08-12 (Actual)

PRIMARY OUTCOMES:
Stress variable | baseline on childbirth first day (before the intervention) .
  The Perceived Stress Scale using 10 items to determine the self-perceived levels of unpredictability, lack of control, and burden during the last month of pregnancy. Responses are rated from 0 (never) to 4 (very often), with higher scores corresponding to higher perceived stress.
Depression variable | baseline on childbirth first day (before the intervention).
  The Edinburgh Postnatal Depression Scale was using 10 items to provide a valuable and efficient way to identify patients at risk of perinatal depression. Each item is scored from 0 to 3, with item scores summed to produce a total The Edinburgh Postnatal Depression Scale was using 10 items to provides a valuable and efficient way to identify patients at risk of perinatal depression. Each item is scored from 0 to 3, with higher scores corresponding to higher depression.
Anxiety variable | baseline on childbirth first day (before the intervention).
  The Beck Anxiety Inventory using 21 items on the scale describes a symptom of anxiety. Responses are rated from 0 (never) to 3 (very often), with higher scores corresponding to higher perceived anxiety.

SECONDARY OUTCOMES:
Stress variable | on childbirth fifth day (after the intervention)
  The Perceived Stress Scale using 10 items to determine the self-perceived levels of unpredictability, lack of control, and burden during the last month of pregnancy. Responses are rated from 0 (never) to 4 (very often), with higher scores corresponding to higher perceived stress.
Depression variable | on childbirth fifth day (after the intervention)
  The Edinburgh Postnatal Depression Scale was using 10 items to provide a valuable and efficient way to identify patients at risk of perinatal depression. Each item is scored from 0 to 3, with item scores summed to produce a total The Edinburgh Postnatal Depression Scale was using 10 items to provides a valuable and efficient way to identify patients at risk of perinatal depression. Each item is scored from 0 to 3, with higher scores corresponding to higher depression.
Anxiety variable | on childbirth fifth day (after the intervention)
  The Beck Anxiety Inventory using 21 items on the scale describes a symptom of anxiety. Responses are rated from 0 (never) to 3 (very often), with higher scores corresponding to higher perceived anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: YUN-FEI PAO, MD, Principal Investigator — Head nurse of research hospital
Locations (1):
- Wan-Lin Pan, Taipei, Taiwan